CLINICAL TRIAL: NCT05021237
Title: A Safety Lead in Single Arm Phase II Study for Image Guided Personalized Ultra-fractionated Stereotactic Adaptive Radiotherapy (PULSAR) for Treatment of Metastatic Cervical Cancer
Brief Title: Personalized Ultra-fractionated Stereotactic Adaptive Radiotherapy for Metastatic Cervical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Elekta Limited (Industry)
Responsible Party: Principal Investigator, Kevin Albuquerque, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0787
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Stage IV Cervical Cancer FIGO 2018; Adenosquamous Carcinoma of Cervix; Cervical Cancer; Metastasis
Keywords: Cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Prospective Therapeutic Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety Lead In (Experimental): An interim safety evaluation will be conducted in a minimum of 10 assessable patients who received at least 3 radiation treatments (pulses) with 90 days follow up after radiation OR who experience a dose-limiting toxicity, as defined below. Patients not meeting these requirements will still count towards the overall trial enrollment target, however, the safety lead-in will continue until 10 fully assessable patients are reached (estimate 17 total patients needed for 40% attrition). These patients initially will be enrolled to the base dose-level of 8.5Gy/fraction.
  Interventions: Radiation: Ultra-fractionated radiation therapy

INTERVENTIONS:
Radiation: Ultra-fractionated radiation therapy — Patients enrolled in this study are planned to receive systemic therapy. Imaging based Ultra-fractionated radiation therapy using a PULSAR technique, which is 5 pulses to gross tumor in pelvis.

SUMMARY:
To improve overall survival in patients with metastatic cervical cancer by loco-regional therapy with personalized ultra-fractionated radiation

DETAILED DESCRIPTION:
The poor outcomes and local morbidity of disease in metastatic cervical cancer, despite evolution in systemic therapy, argues for novel strategies to improve outcome. Improvements in disease control, prevention of morbid local symptoms and even survival have been demonstrated when treating the primary in other cancer types 3,4 Preliminary retrospective data have associated primary site RT with survival benefit in metastatic cervical cancer, but these did not use standardized RT approaches or consider integration with newer systemic therapies28,29. It thus is hypothesized that primary site RT in cervical cancer may achieve similar improvements, but must balance the specific toxicity risks of this disease site and systemic therapy context. Namely, a successful approach must minimize number of treatments to avoid patient inconvenience and systemic therapy interruption, minimize toxicity, and add potential for enhancing systemic disease control. To do this, this study proposes to use PULSAR, implemented by adaptive MRI-guided SAbR in 5 treatments, to deliver primary site cervical RT with ongoing standard systemic therapy. This approaches minimizes treatment visits, doesn't interrupt systemic therapy, uses response-adapted highly conformal RT with advanced image guidance to minimize toxicity risk, and provides potential for improving efficacy of immunotherapy in those receiving it.

ELIGIBILITY:
Inclusion Criteria

1. At least 18 years of age.
2. Ability to understand and the willingness to sign a written informed consent.
3. Newly diagnosed FIGO IVB cervical cancer with radiographic evidence of metastatic disease for whom systemic therapy is standard of care, who are within 6 months of systemic therapy treatment, OR
4. Patients with recurrent/metastatic disease with measurable disease in the pelvis for whom systemic therapy is standard of care and who are within 6 months of initiation of systemic therapy.
5. Patients with brain metastasis are allowed as long as they are clinically stable and/or the mets are treated or are amenable to treatment with radiation and/or surgery.
6. Eastern Cooperative Group (ECOG) performance status of 0-3.
7. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) starting with the first radiation pulse through 90 days after the last fraction of radiation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Medically acceptable birth control (contraceptives) includes:

1) approved hormonal contraceptives (such as birth control pills, patch or ring; Depo-Provera, Implanon), or 2) barrier methods (such as a condom or diaphragm) used with a spermicide (a substance that kills sperm).

A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

  8. Biopsy of primary tumor or recurrent site within 6 months prior to registration

Exclusion Criteria

1. Prior radiation treatment to the pelvis, unless it was for palliation with a total of <=9GY.
2. Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
3. Patients with active Inflammatory Bowel disease or Collagen vascular disease -SLE, scleroderma or on active immunosuppressant (exclusions per PI discretion).
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
5. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
6. Presence of brain metastases that are not amenable to treatment with radiation or surgery, or brain metastasis leading to clinical instability.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only study
Enrollment: 12 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
To determine if image guided ultra-fractionated stereotactic adaptive radiotherapy in metastatic/locally recurrent cervical cancer will improve overall survival outcomes | 2 years
  Overall Survival will be assessed as the percent of patients surviving at each time point. Overall survival is defined as time from diagnosis till death.

SECONDARY OUTCOMES:
To determine the acute and late genitourinary (GU) and gastrointestinal (GI) toxicities | 90 days
  Rates of GU/GI toxicity defined by CTCAE v5 will be measured as acute (≤90 days) and late (> 90 days) up to 1 year from start of radiotherapy
To evaluate the local-regional progression after treatment | 1 year
  The rate of local regional recurrence will be defined as disease recurrence in the treated primary tumor and will measured as a time interval from start of radiation treatment to local progression or death, up to 1 year from start of radiotherapy.

OTHER OUTCOMES:
To determine the treatment response after each pulse of radiation | 1 year
  Change in tumor size on imaging taken during treatment at each fraction (pulse) of radiation for treatments 2-5 and at scheduled imaging up to 1 year from start of radiotherapy
To determine QOL in patients treated with radiation | 1 year
  QOL will be measured using the EORTC QLQ-C30 and EORTC QLQ-CX24
To determine QOL in patients treated with radiation | 1 year
  QOL will be measured using the EORTC QLQ-CX24

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Albuquerque, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States